CLINICAL TRIAL: NCT00728156
Title: Assessment of Platelet-dependent Thrombosis by an ex Vivo Arterial Injury Model: a Placebo Controlled Trial of Clopidogrel as Antiplatelet Therapy in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease
Brief Title: Platelet-dependent Thrombosis: a Placebo-controlled Trial of Antiplatelet Therapy (Clopidogrel)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: British Heart Foundation (Other); University of Newcastle Upon-Tyne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3639a; British Heart Foundation (Other Grant/Funding Number: FS/033/07)
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Artery Disease
Keywords: Type 2 Diabetes mellitus; Coronary artery disease; Platelet dependent thrombogenicity; Aspirin; Clopidogrel; Badimon Chamber
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C (Active Comparator): Patients assigned to clopidogrel in addition to their standard care.(all patients will be on aspirin)We aim to study the effect of clopidogrel as dual antiplatelet therapy in patients with established coronary artery disease and type 2 diabetes. Ninety patients with type 2 diabetes and stable coronary artery disease has been randomly treated with clopidogrel or placebo (45 each) for one week in addition to their standard care (including aspirin,75 mg once daily).
  Interventions: Drug: clopidogrel
- P (Placebo Comparator): Patients assigned to placebo in addition to their standard care.(all patients will be on aspirin).This is a single-centre randomised double-blind placebo-controlled parallel design study, comparing efficacy of clopidogrel versus placebo in patients with T2DM and coronary artery disease. Ninety patients have completed the study. All patients were on their routine medications as per standard practice. After informed consent, participants were randomised to receive either clopidogrel 75mg daily or placebo for 7 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clopidogrel — 75 milligrams, oral, clopidogrel, one tablet daily, for seven days after the baseline chamber study.
  Other Names: Plavix, 75 milligrams; Sanofi Pharma Bristol-Myers Squibb SNC; 174 Avenue de France; F-75013 Paris - France; EU/1/98/069/005a
  Arms: C
Drug: placebo — Placebo: Hydroxy methyl cellulose, similar in weight to the active medication 75 mgs, oral tablets, once a day
  Arms: P

SUMMARY:
Patients with diabetes are more likely to develop furring of their coronary arteries and present with angina and heart attacks. Furthermore, after such an event, they have poorer outcomes (higher rates of death) and survivors are more likely to have recurring symptoms. Using a novel "clotting chamber" the investigators have shown that patients with diabetes are more likely to develop blood clots. This study will look at the role of different blood thinning medications in patients with diabetes. If successful, the investigators will provide evidence to conduct large clinical studies to look at the role of additional blood thinning medication in reducing heart attacks and strokes in patients with diabetes.

DETAILED DESCRIPTION:
The objective of this study is to compare the effect of Clopidogrel on platelet dependent thrombosis in patients with T2DM and CAD with placebo. The Badimon chamber, an ex vivo arterial injury model is used for this purpose. This model simulates the in vivo situation of high shear arterial wall damage and helps to quantify thrombus which is the sum endpoint of all haemostatic abnormalities seen in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM and CAS as defined below:

  * Clinical definitions
  * T2DM: Diagnosed according to the WHO criteria [53].
  * CAD:Presence of any one of the following: Angina plus positive exercise tolerance test, enzyme and/or Q wave positive myocardial infarction, angiographic evidence ( >50% stenosis of one vessel), percutaneous or surgical coronary revascularisation.
* Aged between 18 and 75
* Provided written consent for participation in the trial prior to any study-specific procedures or requirements.

Exclusion Criteria:

* Contraindication to Clopidogrel
* Smoking (current smokers and patients who quit smoking less than six months)
* Malignancy(diagnosed or under investigation)
* Haematological disorders (Anaemia, malignancy, bleeding disorders)
* Women of child-bearing potential
* Use of corticosteroids/other antithrombotic agents(warfarin)
* Chronic liver disease (Cirrhosis, malignancy and patients with more than twice the upper limit of liver function tests)
* Unable to consent.
* Use of other investigational study drugs within 1 year prior to study entry
* Previous participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To compare the effect of Clopidogrel in reduction of thrombogenicity in patients with T2DM and CAD with placebo | seven days

SECONDARY OUTCOMES:
To identify patients (in particular T2DM patients with CAD) resistant to oral antiplatelet therapy | seven days
To characterise features in T2DM patients responsible for increased thrombogenicity | seven days

CONTACTS AND LOCATIONS:
Overall Officials: Azfar G Zaman, MD FRCP, Principal Investigator — Consultant cardiologist and Honoraray Lecturer
Locations (2):
- United Kingdom (2):
  - Newcastle Diabetes Centre, Newcastle General Hospital, Newcastle upon Tyne, Tyne and Wear
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- [Background] Natarajan A, Marshall SM, Worthley SG, Badimon JJ, Zaman AG. The presence of coronary artery disease increases platelet-dependent thrombosis in patients with type 2 diabetes mellitus. J Thromb Haemost. 2008 Dec;6(12):2210-3. doi: 10.1111/j.1538-7836.2008.03176.x. Epub 2008 Oct 1. No abstract available. PMID 18983525
- [Background] Osende JI, Badimon JJ, Fuster V, Herson P, Rabito P, Vidhun R, Zaman A, Rodriguez OJ, Lev EI, Rauch U, Heflt G, Fallon JT, Crandall JP. Blood thrombogenicity in type 2 diabetes mellitus patients is associated with glycemic control. J Am Coll Cardiol. 2001 Nov 1;38(5):1307-12. doi: 10.1016/s0735-1097(01)01555-8. PMID 11691500
- [Background] Shechter M, Merz CN, Paul-Labrador MJ, Kaul S. Blood glucose and platelet-dependent thrombosis in patients with coronary artery disease. J Am Coll Cardiol. 2000 Feb;35(2):300-7. doi: 10.1016/s0735-1097(99)00545-8. PMID 10676673
- [Background] Helft G, Osende JI, Worthley SG, Zaman AG, Rodriguez OJ, Lev EI, Farkouh ME, Fuster V, Badimon JJ, Chesebro JH. Acute antithrombotic effect of a front-loaded regimen of clopidogrel in patients with atherosclerosis on aspirin. Arterioscler Thromb Vasc Biol. 2000 Oct;20(10):2316-21. doi: 10.1161/01.atv.20.10.2316. PMID 11031221
- [Background] Natarajan A, Zaman AG, Marshall SM. Platelet hyperactivity in type 2 diabetes: role of antiplatelet agents. Diab Vasc Dis Res. 2008 Jun;5(2):138-44. doi: 10.3132/dvdr.2008.023. PMID 18537103